CLINICAL TRIAL: NCT06386939
Title: Comparison of Micro- and Macrovascular Disease(s) in People With Type 2 Diabetes, Who Have Moderate to Severe Acanthosis Nigricans vs. Those Who do Not Have Acanthosis Nigricans
Brief Title: Comparison of Micro- and Macrovascular Disease(s) in People With T2D, Who Have Moderate to Severe Acanthosis Nigricans vs. Those Who do Not Have Acanthosis Nigricans
Status: Recruiting | Type: Observational
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Other Study IDs: 01/2024-2025
Record Dates: First submitted 2024-04-20; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus With Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Acanthosis Nigricans: T2DM with Acanthosis Nigricans
- Without Acanthosis Nigricans: T2DM Without Acanthosis Nigricans

SUMMARY:
Hypothesis: Moderate to severe acanthosis nigricans in people with T2D is associated with higher magnitude of complication than people who do not have acanthosis nigricans.

Objectives: To correlate moderate to severe acanthosis nigricans with diabetes complication

Methodology:

T2DM patient will be recruited from endocrine OPD

1. Clinical History and Examination:

1. General Physical Examination: Height, weight, waist circumference, hip circumference, BMI, Blood Pressure, Hand grip. Acanthosis Nigricans.
2. Complications Assessment: Patient will be analysed for:

Micro Vascular

(a) Diabetic retinopathy (i) Mild NPDR (ii) Mod NPDR (iii) Macular Edema / CSME (b) Neuropathy (Mild/Mod/Severe) (c) Chronic Kidney Disease (i) Micro/Macro albumin urea (ii) Increased Creatinine (iii) Decreased eGFR

Macro Vascular

1. Low ABI/PAD
2. CVD-MI/PTCA/CABG/Heart Failure
3. CVS-Stroke/ TIA/Carotid Blockage >50%

DETAILED DESCRIPTION:
The development of type 2 diabetes mellitus (T2DM) as a major public health problem in Asian Indians. Asian Indians develop T2DM at a younger age, and progresses faster than in other ethnic groups. As a result, many diabetes complications are more prevalent and in more advanced stages in Asian countries than in other regions. Asian Indians have one of the highest incidence rates of pre-diabetes and T2DM among all major ethnic groups, and the conversion from pre-diabetes to T2DM occurs more rapidly in this population. According to the Indian Council of Medical Research- India diabetes study (57 117 individuals), the prevalence of prediabetes in all 15 states was 7·3%.

The tendency of Asian Indian to develop T2DM is enhanced by greater insulin resistance, dysglycemia, subclinical inflammation and non-alcoholic fatty liver disease (NAFLD).

Acanthosis nigricans (AN) describes clinically a darkly pigmented thickening skin, which produces epidermal and dermal hyperplasia with orthokeratotic hyperkeratosis and papillomatosis of the stratum spinosum with basal layer hyperpigmentation, in the absence of actual acanthosis and melanocytosis on histologic examination. It is a reactive cutaneous change closely associated with obesity, insulin resistance, and hyperinsulinemia; endocrinopathy; or malignancy, in particular gastrointestinal adenocarcinoma. The prevalence varies, and ethnicity seems an independent factor. Evidence indicates that AN is a useful clinical marker to identify patients susceptible to insulin resistance, the MetS, and type 2 diabetes (T2DM).

This Prospective observational study will be of 12-18 months' duration where 150 T2DM patients from urban areas of Delhi will be randomly screened. The population will be representative of different socio-economic strata of the society. Clinical and dietary profiles, blood pressure and phenotypic markers (acanthosis nigricans, buffalo hump, skin tags: xanthelasma, double chin, arcus, hirsutism and tendon xanthoma), diabetic retinopathy, peripheral arterial disease (PAD), neuropathy, nephropathy HTN, CHF, CT Coronary Angiography, CAD, Arrhythmias, Coronary Calcification, Cerebrovascular Disease, peripheral vascular disease, micro albumin urea, fibro scan and hand grip (average of three values) JAMAR measurement will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM (up to 30 years Duration)
2. Age 20 to 70 years
3. BMI >25 kg/m² to >40 kg/m²
4. Gender- Both (Male & Female)
5. Mild, Moderate and Severe Acanthosis

Exclusion Criteria:

1. Alcoholic with Moderate to Severe.
2. BMI >40 kg/m²
3. Congestive heart disease
4. Positive hepatitis B or hepatitis C, secondary causes of fatty liver (eg. consumption of amiodarone and tamoxifen) and congestive hepatopathy.
5. Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with T2DM visiting Fortis CDOC Hospital will be enrolled in 2 groups cases and controls.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Moderate to Severe Acanthosis Nigricans increases diabetes complications | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — National Diabetes Obesity and Cholesterol Foundation
Locations (1):
- Anoop misra, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No